CLINICAL TRIAL: NCT05274724
Title: Evaluation of the Impact of a Teleconsultation Performed During Ambulance's Displacement on the On-scene Emergency Team's Stay and Patient's Satisfaction
Brief Title: Impact of a Teleconsultation Performed During Ambulance's Displacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 44948821.1.0000.0071
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-03

CONDITIONS: Patients Emergency On-site Care by Mobile Emergency Unit
Keywords: Telemedicine; Ambulance; Transport; Hospital Home Care Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard institutional protocol, without teleconsultation. (Active Comparator): standard will be met according to the current institutional protocol, which does not include teleconsultation. Therefore, the call will be interrupted after guidance from the telemedicine on duty.
  Interventions: Diagnostic Test: No teleconsultation during the ambulance journey
- Teleconsultation during the ambulance journey to the place of care. (Active Comparator): teleconsultation will receive a video call using the free "WhatsApp" application, made by one of the emergency workers of the Telemedicine Center, using an institutional smartphone. The teleconsultation can be done directly to the patient and/or with the companion who made the call. The telemedicine on-duty officer will then assess the condition during the time the ambulance travels. The ambulance team will contact the Telemedicine Center and inform the on-call person when the ambulance geolocation application informs 2 minutes of estimated time of arrival at the place of care. At this point, the on-call doctor will interrupt the teleconsultation and pass the information on to the ambulance team. The video call will be turned off upon arrival of the ambulance team.
  Interventions: Diagnostic Test: Teleconsultation during the ambulance journey

INTERVENTIONS:
Diagnostic Test: No teleconsultation during the ambulance journey — Standard will be met according to the current institutional protocol, which does not include teleconsultation. Therefore, the call will be interrupted after guidance from the telemedicine on duty
  Arms: Standard institutional protocol, without teleconsultation.
Diagnostic Test: Teleconsultation during the ambulance journey — teleconsultation will receive a video call using the free "WhatsApp" application, made by one of the emergency workers of the Telemedicine Center, using an institutional smartphone. The teleconsultation can be done directly to the patient and/or with the companion who made the call. The telemedicine on-duty officer will then assess the condition during the time the ambulance travels. The ambulance team will contact the Telemedicine Center and inform the on-call person when the ambulance geolocation application informs 2 minutes of estimated time of arrival at the place of care. At this point, the on-call doctor will interrupt the teleconsultation and pass the information on to the ambulance team. The video call will be turned off upon arrival of the ambulance team.
  Arms: Teleconsultation during the ambulance journey to the place of care.

SUMMARY:
The establishment of pre-hospital care protocols has shown benefits in the prognosis of numerous acute situations, such as myocardial infarction and stroke, but travel time to the hospital is still a key factor in clinical outcomes. Normally carried out by ambulance, the travel time from the hospital to the place of occurrence is underused. New communication technologies, such as telemedicine, have demonstrated high effectiveness in the management of acute illnesses inside and outside the hospital. Upon arrival at the scene, significant time is spent in properly identifying the problem and obtaining a clinical history. The use of telemedicine is current and simplified in the institution. The hypothesis is that telemedicine contact with companions, family members or the patient himself during the ambulance journey, from the hospital to the place of demand, will be associated with a reduction in the time for carrying out diagnostic hypotheses and for the rescue team to stay on site, as well as greater patient satisfaction. OBJECTIVE: To assess the impact of telemedicine used during the ambulance journey, requests for emergency care, on the time spent by the rescue team at the place of care and on patient satisfaction.

DETAILED DESCRIPTION:
This is a prospective, open, randomized parallel study, with a single telemedicine center and a single emergency service - both at Hospital Israelita Albert Einstein.

Patients who call the emergency service requesting evaluation by the emergency team in their original place will constitute the study population. Patients over 18 years of age and who agree to participate in the study by signing the informed consent will be included. Patients and/or companions without access to the "WhatsApp" application will be excluded, which would make the video call proposed in this experiment impossible.

1. Once the Mobile Emergency Unit is activated by the patient or companion, the ambulance will be sent to the place of care according to institutional protocol.
2. After sending the ambulance, in the case of patients over 18 years of age, the administrative team will transfer the call to the telemedicine emergency team, who will immediately tell the patient about the study and request consent to participate.

   The consent to participate in the study will be recorded in the medical evolution of the telemedicine chart, filled in by the professional of the emergency medical team of the Telemedicine Department who performs the care. This evolution is available in the institutional chart - Cerner Millenium. It will be recorded with the standard phrase: "the participant (PATIENT'S NAME) agreed to participate in the study entitled Assessment of the impact of teleconsultation carried out during ambulance travel on the length of stay of the emergency team at the place of care, whose number CAAE: 44948821.1.0000.0071. All study information will be transmitted only by the medical team professional of the Telemedicine Department to the patient and/or companion who made contact. The information that will be transmitted to the team ambulance, if the patient is randomized to the intervention group, will be: name, age, reason for the call, associated complaints / relevant history data and possible vital signs, relevant background and medications in use. All these data will also be available in the institutional chart. The patient or companion, upon arriving at the HIAE Emergency Care Unit, will fill in the free and informed consent form (delivered by the transport nurse) when there is a clinical opportunity.

   The current care provided by the HIAE Mobile Emergency Unit does not have the participation of a medical team before the arrival of emergency workers at the place of care. Currently, during the entire journey of the ambulance from the base to the place of care for the patient and/or companion, there is no institutional medical evaluation available.

   The study makes it possible to offer evaluation with an institutional medical team also during the displacement of the ambulance. In the two arms proposed for this study, the patient and/or companion will have contact with a professional from the medical team during the displacement of the ambulance, which already adds considerable assistance value.

   The opportunity the investigators found to offer the type of follow-up by the medical team (only by phone versus video and with transmission of information to the team on the move) is immediately after the transfer of the call by the administrative team that received the call from / the patient and / or companion for the Telemedicine Department's emergency team. An objective and standardized conversation is proposed for all cases, following the model below:
   * My name is (PHYSICIAN'S NAME) and I am a telemedicine doctor at Einstein and I will accompany the patient until the ambulance arrives if the patient accept
   * Ambulance will arrive soon
   * The investigators are conducting a simple study to assess whether this conversation of ours can increase the speed of care and increase the speed of transport to the hospital
   * If the patient agree, the investigators will draw which group the patient will participate in (standard care, that is, wait for the ambulance and talk to me to see if I can help with something or telemedicine assistance, where I will call the participant by video, the investigators will talk but I will pass all these data for incoming team). It's simple and it can help.
   * I made the draw and the participant group was (NAME OF THE GROUP DRAWN) The investigators believe that the persistence of the medical team's contact with the patient or companion considerably reduces any type of discomfort for the patient's group to be randomized.
3. If the patient or companion does not agree to participate in the study, the call will be interrupted and the service will proceed normally according to institutional protocol.
4. If the patient or companion agrees to participate in the study, the randomization will be checked and the patient or companion will be informed of the sequence of the study.
5. In view of the short time available between the activation of the mobile emergency unit at Hospital Israelita Albert Einstein and the arrival of the team at the place of care, randomization will be previously established through a randomization application (Randomizer®). The study sample will be analyzed by the application and a 1:1 randomization sequence will be proposed and predetermined. It is noteworthy that the call for pre-hospital care is random. Patients who are included in the study will be randomized according to a pre-established sequence and can be allocated to one of two study groups:

   The. Group I - institution standard: no teleconsultation during ambulance travel to the place of care; B. Group II - teleconsultation: teleconsultation with the patient and/or companion during the ambulance journey to the place of care.
6. Patients allocated to group I - standard will be treated according to the current institutional protocol, which does not include teleconsultation. Therefore, the call will be interrupted after guidance from the telemedicine on duty.
7. Patients allocated to group II - teleconsultation will receive a video call using the free "WhatsApp" application, made by one of the emergency workers of the Telemedicine Center, using an institutional smartphone. The teleconsultation can be done directly to the patient and/or with the companion who made the call. The telemedicine on-duty officer will then assess the condition during the time the ambulance travels. The ambulance team will contact the Telemedicine Center and inform the on-call person when the ambulance geolocation application informs 2 minutes of estimated time of arrival at the place of care. At this point, the on-call doctor will interrupt the teleconsultation and pass the information on to the ambulance team. The video call will be turned off upon arrival of the ambulance team.
8. The nurse of the Mobile Emergency Unit, co-author of the study, when leaving the ambulance after arrival at the place of care, will start timing (available on institutional tablet) and will note two times: length of stay at the place of care (considered until departure ambulance) and transport time to the Morumbi Unit (considered until the ambulance arrives at the emergency room of the Emergency Care Unit of the Morumbi Unit).
9. During the displacement of the ambulance from the place of care to the Morumbi Unit, the nurse of the Mobile Emergency Unit, co-author of the study, will apply the free and informed consent form to all patients or companions. Immediately before arriving at the Morumbi Unit, the same nurse will apply an assessment of service satisfaction through the Net Promoter Score (NPS) printed on a sheet with the question "On a scale of 0 to 10, how much would the participant recommend this service to a friend or family?" An additional unstructured "Why did the participant give this grade?" field will also be populated.
10. The manager of the Mobile Emergency Unit and the Emergency Care Unit are co-authors, participated in the entire preparation of the project and will give their consent in a specific document.

ELIGIBILITY:
Inclusion Criteria:

* Signing the free and informed consent form.

Exclusion Criteria:

* Patients / companions without access to the "WhatsApp" application
* Patients who are not transported to a hospital unit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Length of stay of the emergency team at the point of care | through study completion, an average of 9 months
  Comparison the time spent by emergency team at the point of care, before removing the patient to the hospital, with or without telemedicine consultation.

SECONDARY OUTCOMES:
The time spent by emergency team to perform diagnostic hypotheses | through study completion, an average of 9 months
  Comparison the time spent by emergency team to perform diagnostic hypotheses ,with or without telemedicine consultation.
Total transport time | through study completion, an average of 9 months
  Comparison of total transport time, with or without telemedicine consultation.
Patient or companion satisfaction assessment through Net Promoter Score (NPS) form | through study completion, an average of 9 months
  Comparison the Patient or companion satisfaction assessment through NPS, with or without telemedicine consultation

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo HS Cordioli, MD, Study Director — Telemedicine Department, Hospital Israelita Albert Einstein, Sao Paulo, Brazil
Locations (1):
- Hospital Israelita Abert Einstein, São Paulo, Brazil